CLINICAL TRIAL: NCT03532633
Title: Beobachtungsstudie Zur Versorgung Reif- Und Frühgeborener Mit ausgewählten Mikronährstoffen Wissenschaftliche Untersuchung Bei Minderjährigen
Brief Title: Supply With Micronutrients (Purine and Pyrimidine) in Infants: a Prospective and Observational Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: NEO-MICRO
Record Dates: First submitted 2018-05-09; First posted 2018-05-22 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Prematurity
Keywords: infant; cord; micronutrients; purine; pyrimidine
MeSH Terms: conditions — Premature Birth; Cone-Rod Dystrophies | interventions — Milk, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- 23-27w: preterm infants 23+0-27+6SSW
  Interventions: Procedure: cord blood; Procedure: blood sample infant; Procedure: blood sample mother; Procedure: breast milk
- 28-31w: preterm infants 28+0-31+6SSW
  Interventions: Procedure: cord blood; Procedure: blood sample infant; Procedure: blood sample mother; Procedure: breast milk
- 32-34w: preterm infants 32+0 - 34+6SSW
  Interventions: Procedure: cord blood; Procedure: blood sample infant; Procedure: blood sample mother; Procedure: breast milk
- 35-36w: preterm infants 35+0-36+6 SSW
  Interventions: Procedure: cord blood; Procedure: blood sample infant; Procedure: blood sample mother; Procedure: breast milk
- 37-42w: term infants 37+0-42+6
  Interventions: Procedure: cord blood; Procedure: blood sample infant; Procedure: blood sample mother; Procedure: breast milk

INTERVENTIONS:
Procedure: cord blood — collection of cord blood
Procedure: blood sample infant — collection of remnant of clinically indicated blood sample
Procedure: blood sample mother — collection of remnant of clinically indicated blood sample. If not available blood sample is taken after mother agreed
Procedure: breast milk — collection of breast milk 1/week during neonatal care (maximum 8 weaks)

SUMMARY:
Concentrations of micronutrients (especially purine and pyrimidine) in cord blood, blood of mothers and infants and human milk is studied

DETAILED DESCRIPTION:
Collection of:

1. cord plasma in preterm and term infants.
2. remnants of clinically indicated blood samples of mothers 24 hours before or after birth.
3. remnants of clinically indicated blood samples of preterm and term infants during neonatal care.
4. breast milk once a weak during neonatal care of the infant.

Determination concentrations of micronutrients by mass spectrometry.

Aim is to compare cord plasma concentrations with postnatal plasma concentrations and to measure concentrations in breast milk to determine the actual supply.

Update September 2020:

The results obtained according to the original protocol revealed a serious sample instability when using remnants of clinical blood samples. Remnants can not be used and therefore the protocol had to be changed. A new approval of the Ethics Committee was obtained and is available to the study team. The following changes for sample collection were implemented: an additional blood sample (2.7ml EDTA blood) is taken from the mothers after approval.The blood samples of premature and newborns (max. 3x 0.2 ml) are obtained when a clinically indicated blood sample is taken. In both cases the serum is frozen immediately within one hour after collection.

Due to these changes, the expected end of the study is postponed to 2021.

ELIGIBILITY:
Inclusion Criteria:

* 23+0-42+6 SSW

Exclusion Criteria:

* congenital malformation, genetic disorders
* metabolic disease of the infant
* missing agreement

Ages: 0 Minutes to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: infants and preterm infants
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Concentration of purine and pyrimidine in cord plasma | at birth

SECONDARY OUTCOMES:
Concentration of purine and pyrimidine in neonatal plasma | at times when a clinically indicated blood sample is taken before discharge home from the initial neonatal hospitalization (at a postnatal age of up to 4-5 months at the most in very preterm infants)
Concentration of purine and pyrimidine in breast milk | once a week before discharge home from the initial neonatal hospitalization, maximum 8 weeks
Concentration of purine and pyrimidine in plasma of mothers | 24 hours before and after birth

CONTACTS AND LOCATIONS:
Overall Officials: Axel Franz, Principal Investigator — University Hospital Tuebingen
Locations (1):
- University Children's Hospital Tuebingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No